CLINICAL TRIAL: NCT00874328
Title: A Phase I/II Study of TS-1, Irinotecan and Cisplatin for Patients With Advanced or Metastatic NSLC
Brief Title: A Study of TS-1 Plus Irinotecan and Cisplatin (IP) for Patients With Stage IIIB/IV Non Small Cell Lung Cancer (NSCLC)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Center, Korea (Other Government)
Collaborators: Jeil Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Heung Tae Kim, National Cancer Center, Korea
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCCTS-08-333
Record Dates: First submitted 2008-12-24; First posted 2009-04-02 (Estimated); Last update posted 2010-10-25 (Estimated); Status verified 2010-07

CONDITIONS: Advanced Non-Small Cell Lung Cancer
Keywords: Non small cell lung cancer; Irinotecan plus Cisplatin plus S-1; Phase I/II trial
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Irinotecan; Cisplatin; titanium silicide; S 1 (combination)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- study arm (Experimental): Irinotecan /IV D1 Cisplatin 60mg/m2 iv D1 S-1 bid, P.o. D1 ~ 14 q 3 weeks until maximum 6 cycles
  Interventions: Drug: Irinotecan; Drug: Cisplatin; Drug: TS-1 (S-1)

INTERVENTIONS:
Drug: Irinotecan — Irinotecan iv D1 q 3 weeks until maximum 6 cycles
  Other Names: Campto
Drug: Cisplatin — cisplatin 60mg/m2 iv D1 q 3weeks until maximum 6 cycles
Drug: TS-1 (S-1) — TS-1 po D1~D14 q 3 weeks until maximum 6 cycles
  Other Names: S-1

SUMMARY:
The irinotecan and cisplatin combination showed significant anti-tumor activity. In the first-line setting, the investigators showed that this regimen had significant anti-tumor activity in 47% of chemo-naïve NSCLC patients with 1-year survival rate of 64.2%. Again, the investigators showed that the second-line Irinotecan and cisplatin is an active and well-tolerated regimen in patients with advanced NSCLC pretreated with non-platinum based chemotherapy.

TS-1 (Jeil Pharmaceutical Co.,Ltd, Seoul, Korea) is an oral anticancer drug comprised of tegafur, 5-chloro-2, 4-dihydroxypyridine and potassium oxonate, in a molar ratio of 1:0.4:1. Tegafur is a prodrug that generates 5-fluorouracil (5-FU) in blood via metabolism by liver enzyme, and 5-chloro-2, 4-dihydroxypyridine enhance the serum concentration of 5-FU by the competitive inhibition of dihydropyrimidine dehydrogenase, an enzyme responsible for 5-FU catabolism. Potassium oxonate is also a reversible competitive inhibitor of orotate phosphoribosyl transferase, a phosphoenzyme for 5-FU. Diarrhea induced by 5-FU administration is though to be attributable to the phosphorylation of 5-FU by the enzyme in the gastrointestinal tissue. After oral administration of potassium oxonate, the concentration of potassium in the gastrointestinal tissue is high enough to inhibit the enzyme while the concentration in blood and tumor is reported to be either slight or nil. Because of these mechanism, oral TS-1 administration generates a higher concentration of 5-FU than protracted intravenous infusion of 5-FU given in a dose equimolar to the tegafur in S-1, whereas the incidence of adverse events concerning the GI tract does not increase. In a phase II trial of TS-1 as first-line setting in NSCLC, the response rate was 22% and the median survival time was 10.2 months. As expected, the incidence of severe gastrointestinal adverse events was low, and so was few severe hematologic toxicity. Recently 3-weekly TS-1 plus cisplatin showed activity against NSCLC with a response rate of 32.7% and the safety was acceptable.

DETAILED DESCRIPTION:
The investigators are conducting a phase I/II study to determine the maximum-tolerated dose, the recommended dose, and to evaluate the response rate and toxicity of the TS-1, irinotecan and cisplatin combination in patients with advanced or metastatic NSCLC.

ELIGIBILITY:
Inclusion Criteria:

1. Histologic or cytologic diagnosis of NSCLC, Stage IV or selected stage IIIB (with malignant pleural or pericardial effusion) according to the American Joint Committee on Cancer (AJCC).
2. In phase I, previous chemotherapy including cytotoxic chemotherapy except for irinotecan and cisplatin therapy, targeted therapy and/or radiotherapy is allowed; patients are required to have discontinued previous anti-tumor treatment for at least 4 weeks. Neoadjuvant chemotherapy or adjuvant chemotherapy is allowed and regarded as one-time systemic chemotherapy.
3. In phase II, no prior chemotherapy, radiotherapy or target therapy is allowed. (Prior radiation therapy is allowed as long as the irradiated area is not the only source of measurable disease. Neoadjuvant chemotherapy or adjuvant chemotherapy is not allowed.)
4. Performance status of 0, 1, 2 on the ECOG criteria.
5. At least one uni-dimensionally measurable lesion meeting Response Evaluation Criteria in Solid Tumors (RECIST 2000).
6. Estimated life expectancy of at least 12 weeks.
7. Patient compliance that allows adequate follow-up.
8. Adequate organ function.
9. Metastasis of CNS is not regard to exclusion if the symptom is controlled properly for supportive care including corticosteroid.
10. Informed consent from patient
11. If female: childbearing potential either terminated by surgery, radiation, or menopause, or attenuated by use of an approved contraceptive method (intrauterine device [IUD], birth control pills, or barrier device) during and for 3 months after trial. If male, use of an approved contraceptive method during the study and 3 months afterwards. Females with childbearing potential must have a urine negative hCG test within 7 days prior to the study treatment.

Exclusion Criteria:

1. MI within preceding 6 months or symptomatic heart disease, including unstable angina, congestive heart failure or uncontrolled arrhythmia
2. Serious concomitant infection including post-obstructive pneumonia
3. Second primary malignancy (except in situ carcinoma of the cervix or adequately treated basal cell carcinoma of the skin or prior malignancy treated more than 5 years from the diagnosis without recurrence)
4. Pregnant or nursing women
5. Psychiatric disorder that would preclude compliance.
6. Major surgery other than biopsy within the past two weeks.
7. Patients receiving a concomitant treatment with drugs interacting with S-1 such as flucytosine, phenytoin, or warfarin et al.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2008-10; Primary Completion 2011-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation the Response rate IP plus TS-1(in phase 2) | 1 year

SECONDARY OUTCOMES:
To estimate the time to progression and overall survival | 2 years
Determine MTD (Maximum tolerated dose) in phase I | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Heung Tae Kim, M.D., Principal Investigator — National Cancer Center
Locations (1):
- Asan Medical Center, Seoul, South Korea